CLINICAL TRIAL: NCT05992844
Title: Investigation of the Effect of Kinesthetic Brain Exercise on Fall Risk, Balance and Quality of Life in Hemiplegic Individuals With Stroke
Brief Title: Kinesthetic Brain Exercise in Hemiplegic Individuals With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Betül Taşpınar, PROF. DR., Izmir Democracy University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STROKE-KBE-35
Record Dates: First submitted 2023-07-27; First posted 2023-08-15 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Stroke
Keywords: STROKE; HEMIPLEGIA; COGNITIVE; DYSFUNCTION; EXERCISE
MeSH Terms: conditions — Stroke; Hemiplegia; Motor Activity

STUDY DESIGN:
Intervention Model Description: RANDOMIZED CONTROLLED
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KB Exercises plus Conventional Rehabilitation Group (Experimental): While the participants in the study group will continue the conventional rehabilitation program described below for 3 weeks, lasting 45 minutes on average, 5 sessions a week, they will participate in a total of 9 sessions of kinesthetic brain exercises, 3 sessions a week lasting 30 minutes on average.
  Kinesthetic Brain Exercises Program; The kinesthetic brain exercises program basically consists of 3 phases: warm-up phase, exercise phase and cool-down phase.
  Interventions: Other: KB Exercises Program; Other: Conventional Rehabilitation program
- Conventional Rehabilitation Group (Other): Control Group; Conventional Rehabilitation program; strengthening exercises, balance/gait training, Proprioceptive Neuromuscular Facilitation techniques, neuromuscular electrical stimulation.
  Interventions: Other: Conventional Rehabilitation program

INTERVENTIONS:
Other: KB Exercises Program — Kinesthetic Brain Exercises will carried out for 3 weeks, lasting 45 minutes on average, 5 sessions a week, they will participate in a total of 9 sessions of kinesthetic brain exercises, 3 sessions a week lasting 30 minutes on average.
  Kinesthetic Brain Exercises Program; The kinesthetic brain exercises program basically consists of 3 phases: warm-up phase, exercise phase and cool-down phase.
  Other Names: KINESTHETIC BRAIN EXERCISES
  Arms: KB Exercises plus Conventional Rehabilitation Group
Other: Conventional Rehabilitation program — Conventional Rehabilitation program; strengthening exercises, balance/gait training, Proprioceptive Neuromuscular Facilitation techniques, neuromuscular electrical stimulation.

SUMMARY:
The success of conventional physical therapy in the rehabilitation of stroke patients is demonstrated in the light of studies. In this study, the effects of kinesthetic brain exercises, which is a new exercise approach to be applied together with conventional physiotherapy and rehabilitation, on fall risk, balance, and quality of life will be investigated in hemiplegic individuals who have had a stroke. Thus, it is thought that the effectiveness of kinesthetic brain exercises applied together with conventional physiotherapy and rehabilitation will contribute to the literature for the creation of rehabilitation programs.

DETAILED DESCRIPTION:
Stroke is a clinically defined syndrome characterized by rapidly developing symptoms or signs of cerebral dysfunction with no apparent cause other than vascular causes. Symptoms last more than 24 hours and can lead to death. Findings after stroke; upper and lower extremity motor dysfunctions, spasticity, loss of balance and coordination, walking, swallowing, vision, and communication problems. It has been reported that the disability rate ranges from 13-66% and the disability rate varies between 12-64% due to these functional losses that occur after stroke.

In stroke patients, hemiplegic picture occurs depending on the size and location of the damage in the brain. hemiplegia: It is a paralysis that affects the upper and lower extremities of one side of the body. A decrease in muscle strength, loss of sensation and dysfunction occur on the affected side.

After stroke, the lower extremities are severely affected in hemiplegic individuals. Instability of ankle and knee joints is seen in hemiplegic lower extremities. However, due to instability, the center of gravity shifts towards the unaffected side, which causes balance and coordination disorders. Balance and coordination disorders in hemiplegic individuals cause poor performance in activities and an increased incidence of falls.

Kinesthetic brain exercises: Studies investigating the effects of movement, physical activity and exercises on learning and cognitive development have shown that increased attention span, better focus, better behavioral method, and physical activity that contributes to better learning are supported. Conceptually, brain exercises are expressed by the formula: Physical activity + Brain Activity = Better cognitive function.

Neuroplasticity is the basis of kinesthetic brain exercises. In the light of research, it has been found that the brain is in a state of re-activating the activity that cannot be done by using other ways. In rehabilitation sessions, it is aimed to reconstruct these pathways by transforming daily activities into purposeful exercises. According to Dennison, the founder of kinesthetic brain exercises, brain exercises; It is a combination of physical and mental training with a series of physical movements that activate the whole body in turn, improving the neural connections between the two cerebral hemispheres to enhance learning. Kinesthetic brain training consists of twenty-six simple movements combined with deep breathing. Most of these movements are done diagonally. These diagonal movements result in stimulation and integration of different parts of the brain, especially the corpus callosum, which enables faster and more integrated communication between the two hemispheres in the long run. It is claimed that this situation supports the formation of new neural connections between the two hemispheres of the brain. Drabben et al. In their study, they suggest that brain exercises may be considered a useful physical therapy strategy for older adults, as they can have a positive effect on brain functioning.

The aim of this study is to investigate the effects of kinesthetic brain exercises on lower extremity coordination and balance in hemiplegic individuals who have had a stroke. Thus, it is thought that the effectiveness of kinesthetic brain exercises applied together with conventional physiotherapy and rehabilitation will contribute to the literature for the creation of rehabilitation programs.

Study Hypothesis as follows; Kinesthetic brain exercises have an effect on fall risk, balance and quality of life in hemiplegic individuals who have had a stroke.

ELIGIBILITY:
Inclusion Criteria:

* Being in the 30-60 age range
* Being in the subacute/chronic period (6 months and above).
* Having unsupported sitting balance.
* Having the ability to ambulate with and without support
* Not having botox application for the lower extremities in the last 6 months
* Being at least 3 and above according to the Functional Ambulation Scale
* At least level 3 or higher according to Bruunstrom Lower Extremity Motor Staging.

Exclusion Criteria:

* Having a rheumatological, orthopedic or cardiopulmonary disease that prevents participation in exercises
* Having secondary diseases (MS, Parkinson's, spinal cord injuries, contractures, and post-fracture deformities, etc.)
* Having cognitive, visual, and auditory problems that prevent communication
* Having vestibular system disorders.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
Evaluation of Spasticity | Change from Baseline at 3 weeks
  Upper and lower extremity spasticity status will be evaluated according to the modified Ashworth scale. Spasticity score will be calculated by adding upper extremity spasticity scores of fingers, wrist, elbow and shoulder spasticity scores for upper extremity, and spasticity scores for lower extremity by adding toes, ankle, knee and hip spasticity scores. Higher scores indicate high spasticity.
Brunnstrom Motor Staging | Change from Baseline at 3 weeks
  The Brunnstrom motor assessment is used to evaluate motor function of the hemiplegic side, upper-lower extremities, and hand. According to Brunnstrom, the healing process consists of 6 stages. While the 1st stage is the flaccid stage without isolated movement, the 6th stage is the isolated voluntary movement stage. Only the lower extremity section will be used in this study.
Functional Ambulation Classification (FAS) | Change from Baseline at 3 weeks
  The Functional Ambulation Classification is a widely used ambulation scale that evaluates gait. It is scored between 0 and 5 according to the amount of support the patients receive during walking and consists of 6 categories in total. A score of 0 indicates fully dependent ambulation, while a score of 5 indicates completely independent ambulation.
Activity-Specific Balance Confidence Scale | Change from Baseline at 3 weeks
  It is a self-report form that asks people to evaluate their balance performance during 16 activities determined in the home and outdoor environment. The scale consists of 16 different activities and each item is scored between 0-100. A score of 0 indicates no confidence, and a score of 100 indicates full confidence. The total score is obtained by summing each item score and dividing it by the number of items. A score below 50 indicates a low level, a score between 50-80 indicates a moderate level, and a score above 80 indicates a high level of physical activity.
Timed Sit to Stand Test | Change from Baseline at 3 weeks
  It is a test used to evaluate lower extremity performance and fall risk in stroke patients. During the test, the patient sits on the arm support chair with her back straight and is asked to get up and sit 5 times in quick succession, with her arms crossed on her chest. The elapsed time is recorded in seconds. The patient who cannot stand up unassisted is allowed to get support from the chair and is noted as such. The test is repeated 3 times and the average time is taken. The discrimination cut-off value of this test in stroke individuals is accepted as 12 seconds. If the test takes 15 seconds or more, it is accepted as a risk of repeated falls in elderly individuals.
Timed Up and Go Test | Change from Baseline at 3 weeks
  It is a clinical evaluation test used to evaluate fall risk and dynamic balance in individuals. Patients are asked to sit in an upright position on a chair with an upright back, and with the start command, they are asked to walk 3 meters and return to sit on the chair again. The elapsed time is recorded in seconds. If the patient is walking with an assistive device, he is allowed to walk with an assistive device. The test is repeated 3 times and the average time is recorded. If the test takes more than 14 seconds, it indicates an increased risk of falling in stroke patients.
One Leg Standing Test | Change from Baseline at 3 weeks
  The one leg standing test is used to evaluate static balance and postural control. Patients are asked to stand on one leg. The test is finished when the patient touches the ground when he/she stands up or when he/she stands on one leg for 30 seconds. Both legs are repeated 3 times and the average elapsed time is recorded.
Berg Balance Scale | Change from Baseline at 3 weeks
  Berg balance scale is used to evaluate postural control and fall risk. Berg balance scale consists of 14 items. Each item is scored from 0-4 by observing the performance of the individual. A score of 0 indicates that the patient could not do the activity, and 4 points indicate that she completed the activity independently. According to the Berg balance scale, the highest score that can be obtained is 56, and a score below 45 indicates the risk of falling. A score of 0-20 indicates balance disorder, an acceptable balance between 21-40, and a good balance of 41-56 points.
Assessment of Fall Risk | Change from Baseline at 3 weeks
  This scale consists of 2 sections and 19 risk factors. Major risk factors are given 5 points and minor risk factors are given 1 point. Patients with a score of 5 or more on the scale are considered to have a high risk of falling, and patients with a score of less than 5 are considered to have a low risk of falling.
Stroke-Specific Quality of Life Scale | Change from Baseline at 3 weeks
  This scale consists of 12 fields containing 49 items. These areas are; mobility (6 items), energy (3 items), upper extremity function (5 items), work/production (3 items), temperament (5 items), self-care (5 items), social role (5 items), family role ( It consists of 3 items), vision (3 items), language (5 items), thinking (3 items), and personality traits (3 items). Each fields has a maximum score of 5 and higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Resorlu, Assoc. Prof., Study Chair — Çanakkale 18 March University; Ferruh Taspinar, Prof. Dr., Study Chair — Izmir Democracy University
Locations (1):
- Izmir Democracy University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No